CLINICAL TRIAL: NCT02256085
Title: Treatment of Depersonalization Disorder With Repetitive Transcranial Magnetic Stimulation (rTMS)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: City University of New York, School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 6818
Record Dates: First submitted 2014-08-21; First posted 2014-10-03 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-01

CONDITIONS: Depersonalization Disorder
Keywords: Dissociative; Dissociation; Depersonalization; Depersonalization Disorder; Transcranial Magnetic Stimulation; TMS; DPD; rTMS; Behavioral Symptoms
MeSH Terms: conditions — Depersonalization; Dissociative Disorders; Behavioral Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sham rTMS (Sham Comparator): Daily rTMS with Sham coil
  30 minutes of 1Hz rTMS, 5 days per week, for 6 weeks with Sham (placebo) coil
  Interventions: Device: Daily rTMS with Sham coil
- Active rTMS (Experimental): Daily rTMS with Active coil
  30 minutes of 1Hz rTMS, 5 days per week, for 6 weeks with active coil
  Interventions: Device: Daily rTMS with Active coil
- Open Active rTMS (Experimental): Open Label Daily rTMS with Active coil
  30 minutes of 1Hz rTMS, 5 days per week, for 6 weeks with active coil
  Interventions: Device: Open Label Daily rTMS with Active coil

INTERVENTIONS:
Device: Daily rTMS with Active coil — rTMS produces strong electromagnetic fields (~2Tesla) generated briefly (~1ms) but repetitively (1Hz) applied for 30mins, in five sessions per week for six weeks
  Other Names: Magstim, Magstim Rapid, Magstim Rapid2
  Arms: Active rTMS
Device: Daily rTMS with Sham coil — rTMS produces strong electromagnetic fields (~2Tesla) generated briefly (~1ms) but repetitively (1Hz) applied for 30mins, in five sessions per week for six weeks
  Other Names: Magstim, Magstim Rapid, Magstim Rapid2
  Arms: Sham rTMS
Device: Open Label Daily rTMS with Active coil — rTMS produces strong electromagnetic fields (~2Tesla) generated briefly (~1ms) but repetitively (1Hz) applied for 30mins, in five sessions per week for six weeks
  Other Names: Magstim, Magstim Rapid, Magstim Rapid2
  Arms: Open Active rTMS

SUMMARY:
This is a randomized controlled trial (RCT) on the efficacy of repetitive Transcranial Magnetic Stimulation (rTMS) in the treatment of Depersonalization Disorder (DPD). TMS applies a magnetic field to the brain for a brief period of time. TMS is a procedure that involves 30 minute-long daily sessions every weekday for a series of weeks. The investigators are testing whether TMS can treat Depersonalization Disorder (DPD).

DETAILED DESCRIPTION:
This study is a research trial of an outpatient, non-medication, non-invasive investigational treatment called Transcranial Magnetic Stimulation (TMS). TMS is a noninvasive tool for the study of the human brain that has been approved by the FDA for use in depression, but it is also being investigated as a potential therapeutic agent for other symptoms, such as those seen in Depersonalization Disorder (DPD).

TMS applies a magnetic field to the brain for a brief period of time. TMS is a procedure that involves 30 minute-long daily sessions every weekday for a series of weeks. The investigators are testing whether TMS can treat Depersonalization Disorder (DPD).

In this trial, 32 adult outpatients with DPD, that have been only partially responsive to conventional therapies, will be treated with active or sham low frequency (1 Hz) rTMS applied to the right temporo-parietal junction (TPJ) daily for up to six weeks.

DPD symptoms will be monitored through weekly self-report questionnaires as well clinical ratings with a doctor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients, 18 to 70 years of age.
* Primary diagnosis of Depersonalization Disorder.
* Duration of the index episode of at least a year.
* Patients currently on DPD medication must be at the same stable dose(s) at least 2 months and be to continue at the same dose(s) through the duration of the study.
* Patients must continue to be under the care of their treating psychiatrist who will be writing prescriptions for concomitant medications through the duration of the study.
* Capable and willing to provide informed consent

Exclusion Criteria:

* Individuals diagnosed with current Major Depressive Disorder or Panic Disorder.
* Individuals diagnosed with the following conditions: Bipolar Disorder (lifetime), any Psychotic Disorder (lifetime), History of substance abuse or dependence within the past yea (except nicotine and caffeine).
* Individuals with a neurological disorder including, but not limited to: brain lesion; history of seizures; history of cerebrovascular accident; history of stroke; TIA, cerebral aneurysm, Dementia; Parkinson's Disease; Huntington's chorea; Multiple Sclerosis.
* Increased risk of seizure for any reason, including prior head trauma with loss of consciousness for 5 minutes or more
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease.
* Intracranial implants (e.g. aneurysms clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
* History of treatment with rTMS therapy for any disorder.
* If participating in psychotherapy, must have been in stable treatment for at least three months prior to entry into the study, with no anticipation of change in frequency of therapeutic sessions, or the therapeutic focus over the duration of the rTMS trial.
* Known or suspected pregnancy.
* Women who are breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cambridge Depersonalization Scale (CDS) | Change from baseline after 6 weeks of active rTMS
  The outcome of subjects randomized to active rTMS in phase 1 will be assessed as the change from baseline after 6 weeks of daily rTMS (week 6 assessment). Subjects randomized to receive sham in phase 1 will be assessed at baseline and week 6, but the primary method of assessing improvement will be the change between the baseline and week 12 scores (i.e. after receiving 6 weeks of active rTMS).
  Scale item number: 29 Item score range: Frequency: 0 - 4, Duration: 0-5 Minimum CDS score: 0 Maximum CDS score: 261
  Higher scores indicate the presence of high symptom severity. Decrease in scores from baseline reflects clinical symptom improvement.

SECONDARY OUTCOMES:
Clinical Improvement (assessed by CGI-S) | Change from baseline after 6 weeks of active rTMS
  The outcome of subjects randomized to active rTMS in phase 1 will be assessed as the change from baseline after 6 weeks of daily rTMS (week 6 assessment). Subjects randomized to receive sham in phase 1 will be assessed at baseline and week 6, but the primary method of assessing improvement will be the change between the baseline and week 12 scores (i.e. after receiving 6 weeks of active rTMS).
  Minimum CGI-S score: 1 Maximum CGI-S score: 7
  Higher scores indicate the presence of high symptom severity. Decrease in scores from baseline reflects clinical symptom improvement.
  Patients will be classified as responders with a CGI-S = 1 or 2; and partial responders CGI-S = 3.
  1. = Normal, not at all ill
  2. = Borderline mentally ill
  3. = Mildly ill
  4. = Moderately ill
  5. = Markedly ill
  6. = Severely ill
  7. = Among the most extremely ill patients

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Mantovani, MD, PhD, Principal Investigator — City University of New York; Daniel Javitt, MD, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (2):
- United States (2):
  - Sophie Davis School of Biomedical Education, City University of New York (CUNY), New York, New York
  - New York State Psychiatric Institute, Experimental Therapeutics, New York, New York

REFERENCES:
- [Background] Blanke O, Mohr C, Michel CM, Pascual-Leone A, Brugger P, Seeck M, Landis T, Thut G. Linking out-of-body experience and self processing to mental own-body imagery at the temporoparietal junction. J Neurosci. 2005 Jan 19;25(3):550-7. doi: 10.1523/JNEUROSCI.2612-04.2005. PMID 15659590
- [Background] Chen R, Classen J, Gerloff C, Celnik P, Wassermann EM, Hallett M, Cohen LG. Depression of motor cortex excitability by low-frequency transcranial magnetic stimulation. Neurology. 1997 May;48(5):1398-403. doi: 10.1212/wnl.48.5.1398. PMID 9153480
- [Background] Hunter EC, Baker D, Phillips ML, Sierra M, David AS. Cognitive-behaviour therapy for depersonalisation disorder: an open study. Behav Res Ther. 2005 Sep;43(9):1121-30. doi: 10.1016/j.brat.2004.08.003. PMID 16005701
- [Background] Jimenez-Genchi AM. Repetitive transcranial magnetic stimulation improves depersonalization: a case report. CNS Spectr. 2004 May;9(5):375-6. doi: 10.1017/s1092852900009366. PMID 15115950
- [Background] Sierra M, Phillips ML, Ivin G, Krystal J, David AS. A placebo-controlled, cross-over trial of lamotrigine in depersonalization disorder. J Psychopharmacol. 2003 Mar;17(1):103-5. doi: 10.1177/0269881103017001712. PMID 12680746
- [Background] Simeon D, Guralnik O, Hazlett EA, Spiegel-Cohen J, Hollander E, Buchsbaum MS. Feeling unreal: a PET study of depersonalization disorder. Am J Psychiatry. 2000 Nov;157(11):1782-8. doi: 10.1176/appi.ajp.157.11.1782. PMID 11058475
- [Background] Simeon D, Guralnik O, Schmeidler J, Knutelska M. Fluoxetine therapy in depersonalisation disorder: randomised controlled trial. Br J Psychiatry. 2004 Jul;185:31-6. doi: 10.1192/bjp.185.1.31. PMID 15231553
- [Background] Simeon D, Knutelska M. An open trial of naltrexone in the treatment of depersonalization disorder. J Clin Psychopharmacol. 2005 Jun;25(3):267-70. doi: 10.1097/01.jcp.0000162803.61700.4f. PMID 15876908
- [Background] Simeon D. Depersonalisation disorder: a contemporary overview. CNS Drugs. 2004;18(6):343-54. doi: 10.2165/00023210-200418060-00002. PMID 15089102
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Christopeit M, Simeon D, Urban N, Gowatsky J, Lisanby SH, Mantovani A. Effects of repetitive transcranial magnetic stimulation (rTMS) on specific symptom clusters in depersonalization disorder (DPD). Brain Stimul. 2014 Jan-Feb;7(1):141-3. doi: 10.1016/j.brs.2013.07.006. Epub 2013 Aug 6. No abstract available. PMID 23941986
- See also: Department of Psychiatry, Columbia University Medical Center — http://columbiapsychiatry.org/
- See also: National Institute of Mental Health — http://www.nimh.nih.gov/index.shtml